CLINICAL TRIAL: NCT02990884
Title: Influence of Ultrasonography Guided Ilioinguinal / Iliohipogastric Block in Intraoperative Anesthesia in Children - Randomized Controlled Study
Brief Title: Pediatric Ilioinguinal / Iliohyogogastric Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ERZINCAN UNIVERSITY 6
Record Dates: First submitted 2016-12-04; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Intra-operative Anesthesia and Analgesia Effects
Keywords: Intra-operative anesthesia and analgesia; ilioinguinal / iliohyogogastric nerve block; Pediatric patient
MeSH Terms: conditions — Agnosia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- block and ketamine (Active Comparator): Ilioinguinal / iliohypogastric block after ketamine atropine induction and continued with ketamine only in anesthesia
  Interventions: Drug: ketamine
- ketamine atropine; laryngeal mask (Active Comparator): After ketamine atropine induction, a laryngeal mask was inserted and anesthesia administration was continued with 2 sevoflurane MAC and oxygen / air mixture and applied Ilioinguinal / iliohypogastric block.
  Interventions: Drug: ketamine
- control group (Active Comparator): After ketamine atropine induction, a laryngeal mask was inserted and anesthesia administration was continued with 2 sevoflurane MAC and oxygen / air mixture and Non-block, postoperative analgesia with paracetamol IV
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine

SUMMARY:
Ilioinguinal / iliohyogogastric nerve blocks; It is frequently used for analgesia and anesthesia in inguinal region surgeons. However, 95% of these surgeons are under general anesthesia. aim of this study; Intra-operative anesthesia and analgesia effects of ilioinguinal / iliohyogogastric nerve block supported by ketamine sedation only.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* To undergo elective lower abdominal surgery
* between 2-6 years old

Exclusion Criteria:

* Patients with psychiatric disease
* Patients whose weight is more than 40 kg
* Patients with cardiac-pulmonary-neurological disease
* Patients with bleeding disorder
* Patients with infection or scar on the injection area
* Patients with known allergies to local anesthetics

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
the amount of anesthetic drug which was used | nine month

SECONDARY OUTCOMES:
Postoperative visual analogue scale | nine month

CONTACTS AND LOCATIONS:
Overall Officials: ilke kupeli, Principal Investigator — Erzincan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacroix F. Epidemiology and morbidity of regional anaesthesia in children. Curr Opin Anaesthesiol. 2008 Jun;21(3):345-9. doi: 10.1097/ACO.0b013e3282ffabc5. PMID 18458552
- [Background] Bhattarai BK, Rahman TR, Sah BP, Tuladhar UR. Analgesia after inguinal herniotomy in children: combination of simplified (Single Puncture) ilioinguinal and iliohypogastric nerve blocks and wound infiltration vs. caudal block with 0.25% bupivacaine. Kathmandu Univ Med J (KUMJ). 2005 Jul-Sep;3(3):208-11. PMID 18650577
- [Background] Zanaboni S, Krauss B, Buscaglia R, Montagnini C, Gratarola A, Gualino J, Colombo R, Della Corte F. Changes in respiratory and hemodynamic parameters during low-dose propofol sedation in combination with regional anesthesia for herniorrhaphy and genitourinary surgery in children. Paediatr Anaesth. 2007 Oct;17(10):934-41. doi: 10.1111/j.1460-9592.2007.02299.x. PMID 17767628
- [Background] Abdellatif AA. Ultrasound-guided ilioinguinal/iliohypogastric nerve blocks versus caudal block for postoperative analgesia in children undergoing unilateral groin surgery. Saudi J Anaesth. 2012 Oct-Dec;6(4):367-72. doi: 10.4103/1658-354X.105868. PMID 23493806
- [Background] Seyedhejazi M, Sheikhzadeh D, Adrang Z, Rashed FK. Comparing the analgesic effect of caudal and ilioinguinal iliohypogastric nerve blockade using bupivacaine-clonidine in inguinal surgeries in children 2-7 years old. Afr J Paediatr Surg. 2014 Apr-Jun;11(2):166-9. doi: 10.4103/0189-6725.132821. PMID 24841020
- [Background] Polaner DM, Taenzer AH, Walker BJ, Bosenberg A, Krane EJ, Suresh S, Wolf C, Martin LD. Pediatric Regional Anesthesia Network (PRAN): a multi-institutional study of the use and incidence of complications of pediatric regional anesthesia. Anesth Analg. 2012 Dec;115(6):1353-64. doi: 10.1213/ANE.0b013e31825d9f4b. Epub 2012 Jun 13. PMID 22696610